CLINICAL TRIAL: NCT00309010
Title: Neurophysiology of Task-Specificity of Focal Hand Dystonia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060126; 06-N-0126
Record Dates: First submitted 2006-03-29; First posted 2006-03-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-02-24

CONDITIONS: Focal Dystonia
Keywords: Focal Hand Dystonia; Motor Planning; Transcranial Magnetic Stimulation (TMS); MRI (Magnetic Resonance Imaging); FHD; Writer's Cramp; Healthy Volunteer; HV
MeSH Terms: conditions — Dystonic Disorders; Dystonia, Focal, Task-Specific

SUMMARY:
This study will examine how the brain coordinates movement in patients with focal hand dystonia. Patients with dystonia have muscle spasms that cause uncontrolled twisting and repetitive movement or abnormal postures. In focal dystonia, just one part of the body, such as the hand, neck or face, is involved. This study will use transcranial magnetic stimulation (TMS, see below) to study how the brain plans movement.

Healthy volunteers and patients with focal hand dystonia 18 years of age and older may be eligible for this study. Healthy subjects may participate in one, two or three of the experiments described below. Patients with dystonia may participate in experiments one and three.

Before each experiment, each subject is asked about his/her medical and neurologic history, complete questionnaires and will undergo a brief physical examination.

Experiment 1

* Surface EMG: Small electrodes are taped to the skin over the arm to measure the electrical activity of muscles.
* TMS: A wire coil is held on the subject's scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. During the stimulation, the subject may be asked to tense certain muscles slightly or perform other simple actions. The stimulation may cause a twitch in muscles of the face, arm, or leg, and the subject may hear a click and feel a pulling sensation on the skin under the coil.

Experiment 2 (Two visits.)

* Visit 1: Magnetic resonance imaging (MRI): This test uses a magnetic field and radio waves to obtain images of body tissues and organs. The patient lies on a table that is moved into the scanner (a metal cylinder), wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. The procedure lasts about 90 minutes, during which time the patient will be asked to lie still for up to 30 minutes at a time.
* Visit 2: Surface EMG and TMS

Experiment 3

-Surface EMG and TMS - During the TMS, subjects are asked to respond to shapes on a computer screen by pushing a button or pressing a foot petal.

DETAILED DESCRIPTION:
Objective

Currently, there is no cure for focal hand dystonia (FHD). FHD research has focused predominantly on the motor execution abnormality in the primary motor cortex, while the task-specific nature of FHD has received less attention. Task-specificity suggests that the underlying task-to-motor output relationship is intact for many activities and dysfunctional for an important minority of tasks. The premotor cortex plays a key role in this relationship in health and, likely, plays an equally important role in disordered movement. The goal for this research proposal is to understand the underlying physiology and contribution of the premotor cortex in FHD.

Study population

We intend to study adult patients with FHD and healthy volunteers on an outpatient basis. In a task-specific dystonia of the hand known as writer's cramp, handwriting is abnormal due to posturing and muscle spasm, whereas other tasks done with the affected hand are normal. The disordered relationship between task-to-motor output in FHD is potentially modifiable if the correct target and therapeutic modality are identified.

Design

In a series of three experiments, we propose to use transcranial magnetic stimulation (TMS) to examine the circuitry of the premotor to motor cortex connections in FHD, to interrupt motor planning in FHD, and to define premotor cortex somatotopy. In Experiment 1, TMS will be used to test the hypothesis that there is deficient inhibition from premotor to motor cortex in patients with FHD at rest, during voluntary movement and while maintaining a task-specific position. In Experiment 2, TMS will be used to identify whether there is a somatotopic organization relevant to the inhibitory premotor-motor cortex interaction in healthy volunteers. In Experiment 3, to address the role of motor planning dysfunction in the task-specific nature of FHD, we will use TMS to evaluate the premotor-motor cortex inhibition during a reaction time task.

Outcome measures

The primary outcome measure of Experiment 1 will be change in MEP peak-to-peak amplitude between patients and healthy volunteers at rest and in two motor conditions. In Experiment 2, the primary outcome measure will be the location of the TMS coil for optimizing inhibition from leg premotor cortex to motor cortex compared to the coil location from arm premotor cortex to motor cortex. Finally, in Experiment 3, the primary outcome measure will be the change in reaction time from baseline to the test condition with transient TMS-induced interruption in premotor cortex function.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients:

* Age over 18 years
* Presence of FHD, specifically writer's cramp

Healthy volunteers:

* Age over 18 years
* Absence of dystonia or other neurologic condition

EXCLUSION CRITERIA:

Patients and Healthy volunteers:

* Concurrent medical, surgical, neurologic or psychiatric condition
* Taking medications which include antidepressants, anxiolytics, anticonvulsants, antipsychotics, antiparkinson, hypnotics, stimulants, and/or antihistamines
* Received botulinum toxin injection within 3 months of starting the protocol
* Presence of pacemaker, implanted medical pump, metal plate or metal object in skull or eye
* History of seizure disorder
* For healthy volunteers undergoing MRI, subjects with implanted devices such as pacemakers, medication pumps or defibrillators, metal in the cranium except mouth, intracardiac lines, history of shrapnel injury or any other condition/device that may be contraindicated or prevent the acquisition of MRI and/or current pregnancy
* A serious medical illness which prevents them from lying flat for up to 60 minutes
* Claustrophobia (a fear of tight spaces), which prevents them from lying still in a tight or small space for up to 60 minutes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115
Dates: Start 2006-03-28; Study Completion 2009-02-24

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hallett M. Dystonia: abnormal movements result from loss of inhibition. Adv Neurol. 2004;94:1-9. No abstract available. PMID 14509648
- [Background] Bressman SB. Dystonia genotypes, phenotypes, and classification. Adv Neurol. 2004;94:101-7. No abstract available. PMID 14509661
- [Background] Chen R, Hallett M. Focal dystonia and repetitive motion disorders. Clin Orthop Relat Res. 1998 Jun;(351):102-6. PMID 9646753